CLINICAL TRIAL: NCT06822166
Title: A Single-center, Open-label, Single-sequence, Self-crossover Controlled Phase I Clinical Study Evaluating Methoxyethyl Etomidate Hydrochloride Drug Interactions in Healthy Subjects
Brief Title: Drug Interactions Trial of Methoxyethyl Etomidate Hydrochloride
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ahon Pharmaceutical Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: ET-26-HCL-CP-006
Record Dates: First submitted 2025-01-24; First posted 2025-02-12 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Interaction Drug Food
MeSH Terms: interventions — Rifampin; Fluconazole; Omeprazole; Midazolam

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sequence A (Experimental): rifampicin +ET-26
  Interventions: Drug: rifampicin; Drug: ET-26
- Sequence B (Experimental): Fluconazole+ET-26
  Interventions: Drug: Fluconazole; Drug: ET-26
- Sequence C (Experimental): Omeprazole enteric-coated capsules+midazolam+ET-26
  Interventions: Drug: Omeprazole; Drug: midazolam; Drug: ET-26

INTERVENTIONS:
Drug: rifampicin — rifampicin capsule，600 mg
  Arms: Sequence A
Drug: Fluconazole — Fluconazole capsules: 400 mg for the first dose and 200 mg for the remaining doses
  Arms: Sequence B
Drug: Omeprazole — Omeprazole enteric-coated capsules: 20 mg
  Arms: Sequence C
Drug: midazolam — midazolam injection 0.05 mg/kg was administered intravenously
  Arms: Sequence C
Drug: ET-26 — the dose is 0.8 mg/kg, single dose, Infusion time was 60seconds ± 5seconds

SUMMARY:
Sixty-eight healthy subjects were divided into three sequences: A, B and C. The effects of CYP2C19 inhibitor fluconazole and inducer rifampicin on ET-26-HCl injection were evaluated, and the effects of ET-26-HCl injection on pharmacokinetics of omeprazole and midazolam were evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. healthy adult male and female subjects aged 18-45 years (inclusive);
2. Body weight: body mass index (BMI) between 18.0 and 30.0 kg/m2 (including the cut-off value), with a body weight of at least 50 kg for male subjects and 45 kg for female subjects;
3. The subjects had good communication with the investigators, signed the informed consent form voluntarily, and were able to complete the trial according to the protocol.

Exclusion Criteria:

-

Auxiliary examination:

1. if the results of physical examination, vital signs, 12-lead electrocardiogram, cortisol test, and laboratory tests are abnormal and clinically meaningful;
2. potentially difficult airway;
3. hepatitis B surface antigen, hepatitis C antibody, HIV antibody or syphilis antibody positive;

   Medication history:
4. use of any drugs that inhibit or induce hepatic drug-metabolizing enzymes within 30 days before screening;
5. use of any prescribed medication within 14 days before dosing;
6. use of over-the-counter drugs, Chinese herbal medicines or food supplements such as vitamins and calcium supplements within 7 days before administration;

   History of disease and surgery:
7. any history of clinically severe illness or any disease or condition that the investigator believes may affect the trial results;
8. patients with a history of adrenal insufficiency, adrenal tumors, or hereditary heme biosynthesis disorders;
9. a history of severe cardiovascular disease, including but not limited to a history of organic heart disease, such as heart failure, myocardial infarction, angina, malignant arrhythmia, such as a history of torssion ventricular tachycardia, ventricular tachycardia, long QT syndrome, or symptoms of long QT syndrome and family history;
10. underwent any surgery within 6 months before screening;
11. allergic constitution; Or who, as judged by the investigator, may be allergic to the trial drug or its excipients;

    Living habits:
12. heavy drinking or regular drinking in the 6 months before screening, i.e. drinking more than 14 units of alcohol per week (1 unit =360 mL of beer or 45 mL of 40% spirits or 150 mL of wine); Or with a positive alcohol breath test at baseline;
13. smoked more than 5 cigarettes per day in the 3 months before screening or could not quit smoking during the study;
14. had a history of drug abuse or drug abuse within 3 months before screening; Or the baseline urine drug test was positive;
15. habitual consumption of grapefruit juice or excessive tea, coffee, and/or caffeinated beverages and inability to quit during the trial;

    Others:
16. those who have difficulty in blood collection, can not tolerate venipuncture or arterial blood collection;
17. participated in any other clinical trial within 3 months before screening;
18. vaccinated within 1 month before screening or planned to be vaccinated during the trial period;
19. pregnant or lactating women;
20. childbearing or sperm donation plan during the trial and half a year after the completion of the trial, or do not agree that the subjects and their spouses should take strict contraceptive measures during the trial and half a year after the completion of the trial;
21. had blood loss or donation >400 mL within 3 months before screening, or received blood transfusion within 1 month;
22. subjects with any factors considered by the investigator to be ineligible for the trial.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2023-12-04 (Actual); Primary Completion 2024-01-23 (Actual); Study Completion 2024-01-23 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic Parameter(ET-26/ etomidate acid) | within 1 hour before and 24 hours after the end of ET-26-HCl.from 1 hour before administration of omeprazole enteric-coated capsules until 24 hours after the end of administration.
  Cmax

SECONDARY OUTCOMES:
modified observer's assessment of alert（MOAA/S） score | up to 10 minutes after drug administration.
  The lowest score was 0, indicating full anesthetic sedation, and the highest score was 5, indicating full consciousness.
bispectral index | up to 10 minutes after drug administration.
  BIS values range from 0 to 100, with higher values indicating more wakefulness and lower values indicating more severe cortical inhibition.
Eyelash reflex | up to 2 minutes after drug administration.
  Gently touching the subject's eyelashes with a cotton swab can cause the subject to blink, that is, there is an eyelash reflex. When the eyelash reflex disappears, the patient has entered a state of anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Wei Zhao, Doctor, Principal Investigator — The First Affiliated Hospital of Shandong First Medical University (Qianfoshan Hospital of Shandong Province)
Locations (1):
- The First Affiliated Hospital of Shandong First Medical University (Qianfoshan Hospital of Shandong Province), Jinan, Shandong, China